CLINICAL TRIAL: NCT04861077
Title: Monitoring Breast Cancer Immunotherapy Treatment With Advanced PET/MRI: A Pilot Study
Brief Title: Monitoring Breast Cancer Immunotherapy Treatment With Advanced Positron Emission Tomography Magnetic Resonance Imaging (PET/MRI)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, Director, Advanced Imaging Facility, Director, Division of Molecular Imaging and Therapeutics Professor, Division of Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R21-072; Radiology Research Pilot Award (Other Grant/Funding Number: UAB)
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Breast [18F]FMISO-PET with contrast-enhanced magnetic resonance (MR) (Experimental): The patient will have a plastic peripheral intravenous catheter placed in the arm for administration of 10 millicuries (mCi)/10milliliters (mL) [18F]FMISO (≤ 15 µg/injected dose) followed by an uptake of 120 minutes.
  The injection will be infused nominally over one minute followed by a saline flush. After uptake, the patient will be scanned on the PET/MR for 60 minutes and will receive a contrast injection of gadoteridol during the dynamic sequence of the exam. The patient can be scanned on the PET/CT if the PET/MR is unavailable. During this study patients will be scheduled for up to 3 imaging visits. The first imaging visit will be at baseline prior to starting immunotherapy and is required for study eligibility. If for some reason the patient cannot complete the remaining 2 imaging visits, only one additional imaging visit during the identified times is necessary to remain eligible.
  Interventions: Drug: [18F]FMISO-PET with contrast-enhanced MRI

INTERVENTIONS:
Drug: [18F]FMISO-PET with contrast-enhanced MRI — Triple negative breast cancer patients that are planning to undergo immunotherapy and consent to this study will have 3 imaging visits. Imaging visit 1 will take place before the patients start immunotherapy. Imaging Visit 2 will take place after the patient completes the 1st cycle of immunotherapy and before they start their 2nd cycle. Imaging Visit 3 will take place when the patient completes the 2nd cycle of immunotherapy and before they start the 4th cycle.

SUMMARY:
This clinical study will investigate the utility of Fludeoxyglucose (18F) fluoromisonidazole (FMISO), in patients diagnosed with triple negative breast cancer (stage II-IV disease), to monitor and predict the effect of immunotherapy. This is a parallel imaging study to current treatment strategies and no clinical decisions or outcomes will be based on the imaging. If promising, this data will be used to design larger trials. A total of 20 patients will be recruited for this study. This trial will not designate the participant's treatment plan; they will be eligible based on their treatment plan designated from their oncologist.

DETAILED DESCRIPTION:
Pre-study visit/Consent

This visit will take about 1 hour. Participants will be asked to sign this consent form before any study procedures. Once consented, vital signs will be taken, a blood draw to determine kidney function, and a pregnancy test will be performed for women of childbearing potential. Participants will be asked to fill out an MRI questionnaire and they will be given an additional information sheet on the gadolinium-based contrast agent, Prohance, that the FDA requires for all patients receiving this type of drug. Because the PET/MRI is smaller than most MRI scanners, participants will have a PET/MRI fit test to ensure a proper fit. If eligible for this study, participants will be scheduled for the first PET imaging visit which will occur before they start immunotherapy.

Imaging visits

During this study participants will be scheduled for up to 3 imaging visits. The first imaging visit must be performed before participants start immunotherapy and is necessary for remaining eligible for this study. If, for some reason, the participant misses the following (i.e, 2nd) scheduled imaging visit, they are still eligible to continue in this study as long as they can complete a second imaging visit after finishing the 1st cycle of immunotherapy and before starting the 4th cycle of immunotherapy.

Imaging Visit #1

This visit will take about 4 hours and will take place before the participant starts immunotherapy. No special preparation is required before the study. Upon arrival at the Advanced Imaging Facility (AIF) participants will have a chance to have any remaining questions answered about the procedure. Baseline vital signs, including resting blood pressure, pulse rate, and breathing rate, will be measured and recorded. Women of childbearing potential will have a pregnancy test. An intravenous, plastic catheter will be placed in the arm and participants will be injected with the investigational radioactive drug, [18F]FMISO. Afterwards participants will wait 120 minutes to allow the drug to distribute throughout their body. Participants will then be positioned in the PET/MRI scanner. Based on the PET/MRI fit test, participants will either be positioned face down on their stomach or on their back. Once positioned in the PET/MRI, participants will be imaged for up to 60 minutes during which time they must remain still. During imaging, participants will receive an injection of FDA approved gadolinium-contrast agent called Prohance (gadoteridol) to improve the images.

During any of the imaging visits, if the PET/MRI is unavailable due to scheduling problems or maintenance, participants may be imaged in the PET/CT scanner located in an adjacent room in the AIF. Participants will be scanned for up to 60 minutes. Before or after the PET/CT, but during this visit, participants will receive a separate MRI scan.

When all procedures are complete, the plastic tube will be removed. Unless participants cannot have children because of surgery or other medical reasons, they must agree to use an effective form of birth control for 24 hours after taking the study drug. Effective forms of birth control include birth control pills, patch, intrauterine device (IUD), condom, sponge, diaphragm with spermicide, or avoiding sexual activity that could cause pregnancy. Participants may resume normal activities after that 24-hour waiting period. Participants will be contacted by telephone 48 hours after the procedure to make sure they have not had any type of reaction from the investigational drug.

Imaging Visit #2

The second imaging visit will take about 4 hours and will be scheduled after the participant has finished their 1st cycle of immunotherapy and before they start their 2nd cycle.

No special preparation is required before the study. Upon arrival at the Advanced Imaging Facility (AIF) participants will have a chance to have any remaining questions answered about the procedure. Baseline vital signs, including resting blood pressure, pulse rate, and breathing rate, will be measured and recorded. Women of childbearing potential will have a pregnancy test. An intravenous, plastic catheter will be placed in the arm and participants will be injected with the investigational radioactive drug, [18F]FMISO. Afterwards participants will wait 120 minutes to allow the drug to distribute throughout their body. Participants will then be positioned in the PET/MRI scanner. Based on the PET/MRI fit test, participants will either be positioned face down on their stomach or on their back. Once positioned in the PET/MRI, participants will be imaged for up to 60 minutes during which time they must remain still. During imaging, participants will receive an injection of FDA approved gadolinium-contrast agent called Prohance (gadoteridol) to improve the images.

If participants miss this imaging visit but have completed the 1st imaging visit, they are still eligible to continue in this study if they can complete Imaging Visit #3.

When all procedures are complete, the plastic tube will be removed. Unless participants cannot have children because of surgery or other medical reasons, they must agree to use an effective form of birth control for 24 hours after taking the study drug. Effective forms of birth control include birth control pills, patch, IUD, condom, sponge, diaphragm with spermicide, or avoiding sexual activity that could cause pregnancy. Participants may resume normal activities after that 24-hour waiting period. Participants will be contacted by telephone 48 hours after the procedure to make sure they have not had any type of reaction from the investigational drug.

Imaging Visit #3

The third PET imaging visit will take about 4 hours and will be scheduled after participants finish their 2nd cycle of immunotherapy and before they start their 4th cycle of immunotherapy

No special preparation is required before the study. Upon arrival at the Advanced Imaging Facility (AIF) participants will have a chance to have any remaining questions answered about the procedure. Baseline vital signs, including resting blood pressure, pulse rate, and breathing rate, will be measured and recorded. Women of childbearing potential will have a pregnancy test. An intravenous, plastic catheter will be placed in the arm and participants will be injected with the investigational radioactive drug, [18F]FMISO. Afterwards participants will wait 120 minutes to allow the drug to distribute throughout their body. Participants will then be positioned in the PET/MRI scanner. Based on the PET/MRI fit test, participants will either be positioned face down on their stomach or on their back. Once positioned in the PET/MRI, participants will be imaged for up to 60 minutes during which time they must remain still. During imaging, participants will receive an injection of FDA approved gadolinium-contrast agent called Prohance (gadoteridol) to improve the images.

When all procedures are complete, the plastic tube will be removed. Unless participants cannot have children because of surgery or other medical reasons, they must agree to use an effective form of birth control for 24 hours after taking the study drug. Effective forms of birth control include birth control pills, patch, IUD, condom, sponge, diaphragm with spermicide, or avoiding sexual activity that could cause pregnancy. Participants may resume normal activities after that 24-hour waiting period. Participants will be contacted by telephone 48 hours after the procedure to make sure they have not had any type of reaction from the investigational drug.

The study team will follow participants for up to 5 years or to disease progression by reviewing their medical records including pathology data obtained from surgery to see how they are doing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 years old and ≤ 75 years old
2. Triple negative breast cancer (TNBC) patients (biopsy-proven) stage II-IV eligible
3. >50%Programmed death-ligand 1 (PD-L1) positive
4. Eligible for immunotherapy who are naïve to beginning any immunotherapy treatment
5. May not be pregnant or breastfeeding
6. Subjects must be willing to sign consent
7. Adequate creatinine clearance per institutional guidelines and within 30 days
8. Estimated life expectancy of greater than one year
9. Patients must have one lesion with RECIST measurable disease (greater than 1 cm in diameter, measured from diagnostic breast MRI or staging CT)

Exclusion Criteria:

1. Inability to provide informed consent
2. Weight over 350 lbs., due to the scanner bore size
3. Lactating, known or suspected pregnancy. Women with child-bearing potential must a have a negative serum Human chorionic gonadotropin (β-hCG) pregnancy test within 48 hours or a negative urine β-hCG pregnancy test within 24 hours of each PET imaging study.
4. Contraindication for MRI study (e.g. non-removable metal implants or certain tattoos)
5. Unable to lie still on the imaging table for one (1) hour
6. contraindication for gadolinium-based contrast agent, ProHance (gadoteridol)
7. Have received immunotherapy in the neoadjuvant or adjuvant setting

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Baseline measure of PET standardized uptake value (SUV). | Baseline
  Compare baseline metrics from PET/MRI
Baseline measure of apparent diffusion coefficient (ADC) in mm2/sec from MRI. | Baseline
  Compare baseline metrics from PET/MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Janis O'Malley, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No